CLINICAL TRIAL: NCT06514651
Title: A Phase IA/IB Study to Investigate the Safety, Tolerability, and Pharmacokinetic Characteristics of Intravenous (IV) MAQ-001 as Monotherapy and Combination Immunotherapy in Patients With Advanced Solid Tumors
Brief Title: MAQ-001 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MabQuest SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MQ01
Record Dates: First submitted 2024-06-20; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 1mg/kg of MAQ-001 administered intravenously every 3 weeks
  Interventions: Drug: MAQ-001
- Cohort 2 (Experimental): 3 mg/kg of MAQ-001 administered intravenously every 3 weeks
  Interventions: Drug: MAQ-001
- Cohort 3 (Experimental): 10 mg/kg of MAQ-001 administered intravenously every 3 weeks
  Interventions: Drug: MAQ-001
- Regimen 1 (Experimental): MAQ-001 at 1 mg/kg in combination with ipilimumab at 3 mg/kg administered intravenously every 3 weeks for the first 4 doses, followed by the maintenance phase of MAQ-001 monotherapy administered intravenously at a dose of 3 mg/kg every 3 weeks (q3W)
  Interventions: Drug: MAQ-001; Drug: Ipilimumab
- Regimen 2 (Experimental): MAQ-001 at 3 mg/kg in combination with ipilimumab at 1 mg/kg administered intravenously every 3 weeks for the first 4 doses, followed by the maintenance phase of MAQ-001 monotherapy administered intravenously at a dose of 3 mg/kg every 3 weeks (q3W)
  Interventions: Drug: MAQ-001; Drug: Ipilimumab

INTERVENTIONS:
Drug: MAQ-001 — MAQ-001 is an anti-PD-1 monoclonal antibody that inhibits T cell exhaustion through an alternative mechanism, independent of PD-1/PDL-1 blockade
Drug: Ipilimumab — Ipilimumab is a monoclonal antibody medication that works to activate the immune system by targeting CTLA-4, a protein receptor that downregulates the immune system
  Other Names: Yervoy
  Arms: Regimen 1; Regimen 2

SUMMARY:
The goal of this interventional study is to test a new monoclonal antibody, called MAQ-001, as a potential treatment for certain types of advanced cancers in different organs or compartments, such as skin, lung, kidney, liver, stomach, bowel, the female reproductive system, and hematology lymph node cancers. The main question[s] it aims to answer are:

* the best dose of MAQ-001 that is safe to use alone or in combination with another anti-cancer medicine ipilimumab;
* how MAQ-001 works in the body and how it affects the whole cancer and its cells.

Participants will:

* receive a defined dose of MAQ-001 or MAQ-001 in combination with ipilimumab (depending on rank of enrolment) on day 1 of a 21-day cycle, for a maximum of 2 years.
* receive safety examinations and tumor assessment
* donate blood and other biological materials for safety and pharmacokinetic evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years.
2. Patients who have advanced solid tumors or lymphomas for which an anti-PD-1/PDL-1 has been approved as single agent by the EMA (including but not limited to: melanoma, NSCLC, SCLC, HNSCC, classical HD, primary mediastinal LBCL, urothelial carcinoma, MSI-H cancer, gastric cancer, esophageal cancer, cervical cancer, HCC, merkel, renal cell carcinoma, endometrial cancer, TMB-H cancer, cutaneous SCC, TNBC, unresectable basal cell cancer) with no available approved therapeutic alternatives. In addition, patients with rare tumors for which significant activity of anti-PD1 has been observed (e.g., TLS+ sarcomas, alveolar soft part sarcomas, etc.) may enroll after discussion with the Sponsor.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Histologically/cytologically confirmed diagnosis of a solid tumor malignancy
5. Measurable metastatic disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
6. Life expectancy > 12 weeks
7. Patients who have received prior anti-PD-1, anti-PDL-1, or anti-CTLA-4 therapy or any concurrent chemotherapy, radiotherapy, investigational, biologic, or hormonal therapy for cancer treatment may be eligible to enter the study following a washout period as applicable.
8. Demonstrate adequate organ function
9. Contraception

   * For women: negative pregnancy test for women of child-bearing potential*; must be surgically sterile, postmenopausal, or compliant with an acceptable contraceptive regimen during and for 4 months after the treatment period. Abstinence is not considered an adequate contraceptive regimen.
   * For men: must be surgically sterile, or compliant with a contraceptive regimen during and for a minimum of 4 months after the treatment period.
10. Adequate knowledge in speaking and reading local language. * A woman is considered of childbearing potential (WOCBP), i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

Exclusion Criteria:

1. Patients have a known uncontrolled central nervous system (CNS) metastases and/or carcinomatous meningitis or untreated CNS metastatic disease, leptomeningeal disease, or cord compression.
2. Patients have a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
3. Patients have a known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid (HCV RNA) (qualitative) is detected).
4. Patients have participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of study drug.
5. Patients have received prior anti-cancer therapy (chemotherapy, targeted therapies, radiotherapy, or immunotherapy) within 21 days, or less than 5 times the half-life of the most recent therapy prior to study Day 1, whichever is shorter.
6. Patients have not recovered adequately (≤ Grade 1) from AEs and/or complications from any major surgery prior to starting therapy.
7. Patients who have an active autoimmune disease requiring systemic treatment within the past 3 months or have a documented history of clinically severe autoimmune disease that requires systemic steroids or immunosuppressive agents.
8. Patients have a history of organ transplant that requires use of immune suppressive agents.
9. Patients have an active malignancy not related to the current diagnosed malignancy.
10. Patients must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy, including but not limited to grade ≥2 myocarditis, grade ≥3 pneumonitis, or grade ≥3 toxicities not listed above.
11. All AEs while receiving prior immunotherapy must have completely resolved or resolved to Grade 1 prior to screening for this study.
12. Patients taking steroids at a dose >10 mg prednisone equivalent daily, or any other immunosuppressive drugs within 28 days prior to the first dose of MAQ-001. However, patients are allowed to use topical or inhaled glucocorticoids and adrenal glucocorticoids replacement therapy at an effective dose equivalent to ≤ 10 mg/day of prednisone.
13. Uncontrolled intercurrent illness, that would limit compliance with study requirements, substantially increase the risk of incurring AEs or compromise the ability of the subject to give written informed consent.
14. Any condition that, in the opinion of the investigator, would interfere with the evaluation of the investigational product or interpretation of the patient's safety or study results, or not suitable for inclusion as judged by the investigator.
15. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions, and requirements.
16. Patients had cerebrovascular accident, myocardial infarction, unstable angina, poorly controlled arrhythmia occurring within 6 months of enrollment.
17. Patients have cardiac insufficiency of Grade III or IV according to the New York Heart Association (NYHA) classification.
18. Patients have interstitial pneumonitis, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, and/or severely impaired lung function, that may interfere with the detection and management of suspected MAQ-001-related pulmonary toxicity.
19. Administration of live vaccines within 28 days prior to the first dose. Patients may receive inactivated viral vaccines for seasonal influenza and 2019-nCoV vaccines but may not receive live attenuated influenza vaccines via the intranasal route.
20. Patients had a major surgery within 28 days prior to the first dose of investigational product. A major surgery is defined as a surgery that takes at least 3 weeks of postoperative recovery before receiving treatment in this study.
21. Patients have known hypersensitivity or contraindication to anti-PDL1.
22. For patients in Phase IB: known hypersensitivity or contraindication to ipilimumab.
23. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) in monotherapy and in combination with ipilimumab at the end of Phase IA and IB, respectively | up to 2 years
  Number and percentage of subjects experiencing Treatment Emergent Adverse Event (TEAE), serious TEAE, TEAE related to investigational products and serious TEAE related to investigational products will be described as well as the number and percentage of events by dose level and overall
Maximum Administered Dose (MAD) in monotherapy and in combination with ipilimumab at the end of Phase IA and IB, respectively | up to 2 years
  Number and percentage of subjects experiencing Treatment Emergent Adverse Event (TEAE), serious TEAE, TEAE related to investigational products and serious TEAE related to investigational products will be described as well as the number and percentage of events by dose level and overall
Incidence and severity of treatment-emergent adverse events (TEAEs) throughout the observation period | First 21-day treatment cycle
  Number and percentage of subjects experiencing Treatment Emergent Adverse Event (TEAE), TEAE related to investigational products products will be described as well as the number and percentage of events by dose level and overall
Incidence and severity of treatment-emergent serious adverse events (TESAEs) throughout the observation period | First 21-day treatment cycle
  Number and percentage of subjects experiencing serious Treatment Emergent Adverse Event (TEAE), serious TEAE related to investigational products will be described as well as the number and percentage of events by dose level and overall
Incidence and severity of Dose Limiting Toxicity (DLT) during the first 21-day treatment cycle | First 21-day treatment cycle
  number and percentage at each dose level and number and percentage of patients who will have developed a DLT in the first 21 days in each dose level

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Léon Bérard, Lyon
  - Institut Gustave Roussy, Paris
  - Centre Eugene Marquis, Rennes
  - Oncopole Claudius Regaud Toulouse, Toulouse